CLINICAL TRIAL: NCT00590304
Title: Asthma in the Delta Region of Arkansas: Characterization of Disease and Impact of Environmental Factors
Acronym: ADRA
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 53054
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Asthma, Children, Rural Population, Morbidity, Endotoxin
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Optional buccal swab samples will be obtained from participants. This is done by touching the inside of the participant's cheek to collect a sample of the cells in his/her mouth with a cotton swab type applicator.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EU, LV, MA, EL, DU: The population will consist of 120 English-speaking participants ages 4-17 years from four rural schools with physician-diagnosed asthma or symptoms of asthma in the previous 12 months. As of June 2008, an additional rural school has been added to the population criteria, making a total of five rural schools.

SUMMARY:
The purpose of the study is to evaluate asthma and examine the homes of children with asthma living in rural areas of the state. This study is being done to give investigators more information about the presence of allergens and endotoxin in the homes of children with asthma living in the delta region of Arkansas.

DETAILED DESCRIPTION:
Asthma is the most common chronic disease of children and disproportionately affects minority and low-income children. Current pediatric asthma research in this high-risk group focuses on children living in inner-city environments. Low-income, minority children with asthma from non-urban locales have not been studied extensively. The specific aims of the study will examine the impact of home environmental exposure to endotoxin on asthma severity and atopy status in the rural setting among predominately African American, low-income asthmatics. This study will answer several research questions. The first question involves the relationship between asthma severity and exposure to endotoxin among rural children at high risk for increased morbidity and mortality. Second, the relationship between atopy and endotoxin exposure has been the subject of recent debates among asthma researchers. The hygiene hypothesis suggest that the recent rise in atopic disease in Westernized societies is due to decreased microbial burden. Last data on atopy and aeroallergen exposure among high-risk rural asthmatics will be critical in the design and implementation of future intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* English speaking participants aged 4-17 years from four rural schools with physician diagnosed asthma or symptoms of asthma in the previous 12 months (coughing, wheezing, chest tightness, shortness of breath) (per parental or legal guardian report) and current taking prescribed medications for asthma such as inhalers, syrup or breathing machine.

Exclusion Criteria:

* Children with significant underlying respiratory disease other than asthma (such as cystic fibrosis) or significant co-morbid conditions such as severe developmental delay or cerebral palsy will be excluded from the study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be children with asthma, ages 4-17 years from the Mississippi Delta region. The Mississippi Delta has been identified as one of the poorest, medically-underserved regions of the United States, and includes the geographic regions of Arkansas, Louisiana and Mississippi that are contiguous with the Mississippi River. Participants for the study will be recruited from Eudora, Lake Village, Marvell and Elaine public school districts. Since June 2008, the Dumas Public School District has been added in the recruitment. These districts are located in the Delta region of Arkansas where more than one-third of families with children 5-17 years are below the 2000 poverty line (Census bureau). Students in these school districts are predominately of a miniority population.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Asthma morbidity data will be analyzed to examine relationships between home environment factors and morbidity outcomes such as symptom frequency, medication use, healthcare utilizations and decreased activity. | Three years

SECONDARY OUTCOMES:
The study will yield preliminary and feasibility data critical for designing future large-scale asthma studies among high-risk populations. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual data.

REFERENCES:
- [Background] Perry TT, Vargas PA, McCracken A, Jones SM. Underdiagnosed and uncontrolled asthma: findings in rural schoolchildren from the Delta region of Arkansas. Ann Allergy Asthma Immunol. 2008 Oct;101(4):375-81. doi: 10.1016/S1081-1206(10)60313-4. PMID 18939725
- [Result] Pesek R, PA V, Jones S, McCracken A, Perry TT. Pediatric asthma diagnosis and morbidity in urban and rural Arkansas. J Allergy Clin Immunol 2009;123:S210.
- [Result] Haynes A, Vargas PA, Watkins D, Brown R, McCracken A, Jones S. Allergen exposure and home characteristics of high risk rural children with asthma. J Allergy Clin Immunol 2008;121:S231.
- [Derived] Coleman AT, Rettiganti M, Bai S, Brown RH, Perry TT. Mouse and cockroach exposure in rural Arkansas Delta region homes. Ann Allergy Asthma Immunol. 2014 Mar;112(3):256-60. doi: 10.1016/j.anai.2014.01.002. Epub 2014 Jan 31. PMID 24491312
- [Derived] Perry TT, Rettiganti M, Brown RH, Nick TG, Jones SM. Uncontrolled asthma and factors related to morbidity in an impoverished, rural environment. Ann Allergy Asthma Immunol. 2012 Apr;108(4):254-9. doi: 10.1016/j.anai.2012.01.017. Epub 2012 Feb 15. PMID 22469445